CLINICAL TRIAL: NCT04517604
Title: Feasibility of a Combined Neuromodulation and Yoga Intervention for Veterans With Mild Traumatic Brain Injury and Chronic Pain
Brief Title: Neuromodulation and Yoga for Mild Traumatic Brain Injury and Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N3611-P; I21RX003611 (NIH)
Record Dates: First submitted 2020-07-17; First posted 2020-08-18 (Actual); Results first posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Mild Traumatic Brain Injury; Chronic Pain
Keywords: traumatic brain injury; concussion; chronic pain; pain; neuromodulation; transcranial magnetic stimulation; intermittent theta burst stimulation; yoga
MeSH Terms: conditions — Brain Concussion; Chronic Pain; Brain Injuries, Traumatic; Pain

STUDY DESIGN:
Intervention Model Description: Intermittent Theta Burst Stimulation (iTBS) in combination with Love Your Brain Yoga Program. 6 weekly sessions of iTBS given prior to small group yoga.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- iTBS+yoga (Experimental): Participants will receive 6 sessions of intermittent theta burst stimulation (iTBS) and the LoveYourBrain Yoga program. The LoveYourBrain Yoga program was specifically designed for people with TBI.
  Interventions: Device: Magventure MagProx100 with MagOption

INTERVENTIONS:
Device: Magventure MagProx100 with MagOption — The Magventure C-B60 butterfly coil will be used for single-pulse TMS to determine motor threshold. iTBS will be delivered utilizing the MagVentrure MagPro X100 with MagOption stimulator that includes active and placebo coils (C-B65 Butterfly coils) or active-only Cool-B65 Butterfly (figure 8) coil. Only the active setting will be used.

SUMMARY:
The objectives of this VA SPiRE application are to develop a combined neuromodulation and yoga (iTBS+yoga) intervention for Veterans with mild traumatic brain injury (mTBI) and chronic pain, assess the intervention's feasibility and acceptability, and to gather preliminary clinical outcome data on quality of life, function and pain that will guide future studies. This SPiRE project will directly benefit Veterans and VA Services by developing a new, non-pharmacological neurorehabilitation treatment for Veterans with mTBI and chronic pain in need of non-opioid treatment options. Neuromodulation is now offered at 30 VA hospitals and yoga is among the complementary and integrative health programs being rolled out as a part of VAs Whole Health implementation efforts. Thus, should iTBS+yoga ultimately prove to be efficacious, VA facilities will be well-poised to offer this treatment. A novel, activity-based, non-pharmacological treatment for Veterans with mTBI and chronic pain is of great need given the high prevalence of chronic pain.

DETAILED DESCRIPTION:
Over 340,000 people have incurred a mild traumatic brain injury (mTBI) as a result of the military conflicts in Iraq and Afghanistan. mTBI leads to a host of poor rehabilitation outcomes including impairments in cognition, physical health, and psychological health. These impairments among people with TBI lead to poor quality of life (QOL). Worsening this clinical picture, the prevalence of chronic pain is estimated to be 51.5% among civilians with TBI and 43.1-70% among Veterans with TBI. Opioids are used for treating chronic pain including among people with TBI. Thus, given the ongoing opioid epidemic in the United States, it is very timely to develop alter-native, non-pharmacologic treatments for chronic pain among Veterans with mTBI. Yoga is a promising activity-based intervention for TBI and chronic pain. Yoga is an activity generally comprised of breathing exercises, gentle stretching, and meditation. Neuromodulation through transcranial magnetic stimulation (TMS) is a prom-ising non-invasive, non-pharmacological treatment for TBI and chronic pain. Intermittent theta burst stimulation (iTBS) is a type of patterned, excitatory TMS. iTBS can induce a window of neuroplasticity, making it ideally suited to boost the effects of treatments provided after it. Thus, iTBS shows promise to prime the brain for combined interventions and may magnify the impacts that these interventions would have when used alone, in order to boost outcomes. The purpose of this SPiRE project is to develop a novel, combined neuromodulation and yoga neurorehabilitation intervention for Veterans with mTBI and chronic pain, and to examine the intervention's feasibility and acceptability. Using an existing, evidence-based, yoga program created specifically for people with TBI (LoveYourBrain Yoga), the investigators will first develop a neurorehabilitation intervention that combines iTBS with yoga (iTBS+yoga), and then collect pilot data about its feasibility and acceptability. Aim 1 will develop a novel, combined iTBS+yoga neurorehabilitation intervention for Veterans with mTBI and chronic pain. Aim 2 will examine the feasibility and acceptability of the iTBS+yoga intervention for Veterans with mTBI and chronic pain. Aim 3 will gather preliminary data to provide the foundation for sample size and power considerations for a future clinical trial to examine the effectiveness of iTBS+yoga on Veterans' quality of life, function and pain out-comes. The combined intervention will be provided in small group settings once a week for 6 weeks. iTBS will be administered immediately prior to the LoveYourBrain Yoga session. Emphasizing National Institute of Neuro-logical Disorders and Stroke (NINDS) Traumatic Brain Injury Common Data Elements (TBI CDEs), the investigators will collect preliminary outcome data related to quality of life, function and pain to inform a future Merit application, should the intervention prove feasible. This SPiRE project will directly benefit Veterans and VA Services by developing a new, non-pharmacological neurorehabilitation treatment for Veterans with mTBI and chronic pain in need of non-opioid treatment options. TMS is now offered at 30 VA hospitals nationwide for treatment-resistant depression, and yoga is among the complementary and integrative health programs being rolled out as a part of VAs nation-wide Whole Health implementation efforts, with classes offered through VA service lines such as recreational therapy. Therefore, should iTBS+yoga ultimately prove to be efficacious and effective, VA facilities will be well-poised to offer this treatment. A novel, activity-based, non-pharmacological treatment for Veterans with mTBI and chronic pain is of great need given the high prevalence of chronic pain, increased risk of opioid therapy, and increased risk of developing opioid use disorders.

ELIGIBILITY:
Inclusion Criteria:

* 22+ years of age
* Can read and speak English
* Perceive themselves as able to participate in gentle physical movements and cleared by study physician to do so.
* mTBI Criteria: Symptom Attribution and Classification (SACA) criteria for mTBI (without requirement of clinical neuropsychological impairment)
* Chronic pain: pain that persists for >6 months and is of moderate to severe intensity with a score of >5 on specific items on the Brief Pain Inventory (BPI)
* Fully vaccinated against COVID-19 prior to study participation

Exclusion Criteria:

* Contraindications to iTBS/TMS (e.g. epilepsy, history of anoxic brain injury or heart disease)
* Contraindications to MRI (e.g., claustrophobia, ferromagnetic metal implants)
* Pain believed to be associated with cardiac or ischemic conditions
* Active seizure disorder, or if they are taking psychostimulants (e.g. amphetamines), anticholinergics or other medications that may increase their risk of having seizures
* History of moderate to severe TBI
* History of or current psychosis not due to an external cause (e.g., due to illicit drug use)
* Are pregnant or nursing
* Within 12 weeks of a major surgery/operation
* Have questionably valid test profiles

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy A Herrold, PhD BA, Principal Investigator — Edward Hines Jr. VA Hospital, Hines, IL
Locations (1):
- Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified data set will be created and shared.Final data sets will be made available as per Hines VA Hospital local policy for long term storage and access until enterprise-level resources become available. These data will be available upon request by researchers and scientists in accordance with federal guidelines and Hines local policy.
  The data provided will be sufficient for anyone to perform analogous or supplemental analyses that would permit validation of the analysis and results. The sharing of data will enable others to evaluate the data and to validate and interpret the data independently. In order to insure that replication is possible and transparency, statistical code complementary to datasets will be made available through the Federal Interagency Traumatic Brain Injury Research Informatics System.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: After primary publication of study data.
Access Criteria: These data will be available upon request by researchers and scientists in accordance with federal guidelines and Hines local policy.

REFERENCES:
- [Derived] Krese KA, Donnelly KZ, Etingen B, Bender Pape TL, Chaudhuri S, Aaronson AL, Shah RP, Bhaumik DK, Billups A, Bedo S, Wanicek-Squeo MT, Bobra S, Herrold AA. Feasibility of a Combined Neuromodulation and Yoga Intervention for Mild Traumatic Brain Injury and Chronic Pain: Protocol for an Open-label Pilot Trial. JMIR Res Protoc. 2022 Jun 15;11(6):e37836. doi: 10.2196/37836. PMID 35704372

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited treatment-seeking Veterans from Edward Hines Jr., VA Hospital Recruitment Period: 6/2021 to 6/2023 Types of Location: Suburban VA Hospital and associated relevant clinics such as the Polytrauma/TBI clinic.
Pre-assignment Details: Participants were screened over the phone with a delimited set of measures but more in-depth screening for full eligibility criteria occurred after consent/enrollment. Thus, only enrolled participants meeting full eligibility criteria were allowed to move forward and assigned to receive the treatment intervention.
Period: Overall Study
Arm/Group | iTBS+Yoga
Started | 19
Completed | 10
Not Completed | 9

BASELINE CHARACTERISTICS:
Population: 19 participants enrolled, 14 initiated iTBS+yoga sessions, and 10 completed all sessions
Groups:
- Open Label iTBS+Yoga: All patients received individual approximately 3-minute iTBS session followed by a 90-minute group LoveYourBrain yoga session. iTBS+yoga sessions occurred once a week for 6 weeks.
Arm/Group | Open Label iTBS+Yoga
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 43.1 [24 to 64]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: cisgender men | 13
  Gender: cisgender women | 5
  Gender: transgender men | 1
  Gender: transgender women | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 7
  White | 9
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19
Brief Pain Inventory - Pain Severity [Mean (Standard Deviation); unit: units on a scale] — 4 main items and each item is scored on a scale of 0 to 10 with 0 meaning no pain, and 10 meaning pain as bad as you can imagine. Minimum (best) score for all 4 items would be 0 and maximum (worst) score would be 40. Population: All participants that completed baseline assessments are included which is an n=14.
  units on a scale
    number analyzed (Participants) | 14
    (all) | 5.59 (1.36)
Brief Pain Inventory - Pain Interference [Mean (Standard Deviation); unit: units on a scale] — 7 main items and each item is scored on a scale of 0 to 10 with 0 meaning does not interfere, and 10 meaning completely interferes. Minimum (best) score for all 7 items would be 0 and maximum (worst) score would be 70. Population: All participants who completed baseline measures are included which is an n=14.
  units on a scale
    number analyzed (Participants) | 14
    (all) | 4.24 (2.80)
Mayo-Portland Adaptability Inventory (MPAI-4) - Total [Mean (Standard Deviation); unit: T-Score] — Mayo-Portland Adaptability Inventory (MPAI-4) Total T-Score. The Total raw score is converted to a T-score using a national sample conversion chart provided in the MPAI-4 manual. Mean = 50, Standard deviation = 10. Higher scores represent worse function and lower scores indicate better function. Population: All participants who participated in baseline assessments are reported which is an n=14.
  T-Score
    number analyzed (Participants) | 14
    (all) | 39.3 (9.03)
Mayo-Portland Adaptability Inventory (MPAI-4) - Ability [Mean (Standard Deviation); unit: T-Score] — Mayo-Portland Adaptability Inventory (MPAI-4) Ability Index Subscale T-Score. The Ability Index Subscale raw score is converted to a T-score using a national sample conversion chart provided in the MPAI-4 manual. Mean = 50, Standard deviation = 10. Higher scores represent worse function and lower scores indicate better function. Population: All participants who completed baseline assessments are included which is an n=14.
  T-Score
    number analyzed (Participants) | 14
    (all) | 39.7 (9.87)
Mayo-Portland Adaptability Inventory (MPAI-4) - Participation [Mean (Standard Deviation); unit: T-Score] — Mayo-Portland Adaptability Inventory (MPAI-4) Participation Index Subscale T-Score. The Participation Index Subscale raw score is converted to a T-score using a national sample conversion chart provided in the MPAI-4 manual. Mean = 50, Standard deviation = 10. Higher scores represent worse function and lower scores indicate better function. Population: All participants who completed baseline assessments which is an n=14 are included.
  T-Score
    number analyzed (Participants) | 14
    (all) | 31.5 (10.6)
Mayo-Portland Adaptability Inventory (MPAI-4) - Adjustment [Mean (Standard Deviation); unit: T-Score] — Mayo-Portland Adaptability Inventory (MPAI-4) Adjustment Index Subscale T-Score. The Adjustment Index Subscale raw score is converted to a T-score using a national sample conversion chart provided in the MPAI-4 manual. Mean = 50, Standard deviation = 10. Higher scores represent worse function and lower scores indicate better function. Population: All participants that completed baseline assessments are included which is an n=14.
  T-Score
    number analyzed (Participants) | 14
    (all) | 46.7 (7.49)

OUTCOME MEASURES:

1. Primary Outcome: Session Completion Rate
Description: For feasibility, we will track the number of iTBS+yoga sessions completed and compute completion percentage rates for each participant as a metric of feasibility.
Time Frame: Endpoint - after last iTBS+yoga session, approximately 6 weeks
Population: 14 participants initiated iTBS+yoga treatment sessions and could possibly complete 6 total number of intervention sessions. Thus total number of possible sessions is 14 x 6 = 84
Measure: Count of Units; unit: number of sessions
Units Other Than Participants: number of sessions
Arm/Group | iTBS+Yoga
Number analyzed (Participants) | 14
Number analyzed (number of sessions) | 84
number of sessions | 60

2. Secondary Outcome: Mayo-Portland Adaptability Index - Total
Description: The Mayo-Portland Adaptability Index is a TBI Common Data Element assessment of function and participation. It includes 35 items each scored on a scale of 0 to 4, with 0 meaning no problems (better), and 4 meaning severe problems (worse). Minimum (best) score would be 0 and maximum (worst) score would be 140.
Time Frame: Endpoint (after last iTBS+yoga treatment, approximately 6 weeks)
Population: Analysis completed on the 10 iTBS+yoga treatment completers
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label iTBS+Yoga
Number analyzed (Participants) | 10
score on a scale | 35.2 (17.4)
Statistical Analysis 1: Comparison: Open Label iTBS+Yoga; Test type: Superiority; p = .343, Mixed Models Analysis — no adjustment for multiple comparisons as was a pilot; Mean Difference (Final Values) = -5.02, 95% CI 2-sided [-16.52 to 6.47], Standard Deviation 4.984

3. Secondary Outcome: Brief Pain Inventory - Pain Severity
Description: The Brief Pain Inventory is a self-report measure of pain symptoms throughout the body. It has 4 main items and each item is scored on a scale of 0 to 10 with 0 meaning no pain (better), and 10 meaning pain as bad as you can imagine (worse). Minimum (best) score would be 0 and maximum (worst) score would be 40.
Time Frame: Endpoint (after last iTBS+yoga treatment, approximately 6 weeks)
Population: Analysis completed on the 10 iTBS+yoga treatment completers
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label iTBS+Yoga
Number analyzed (Participants) | 10
score on a scale | 3.7 (1.5)
Statistical Analysis 1: Comparison: Open Label iTBS+Yoga; This was an open-label, single group study using a within subject design. We compared pre-treatment values to post-treatment values; Test type: Superiority — This was a pilot study funded under a pilot funding mechanism which specifically did not require a power analysis; p = .0026, Mixed Models Analysis — no test for multiple comparisons as this was a pilot study; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-2.63 to -.77], Standard Deviation .42

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Safety data on safety indicators was collected at each iTBS session including the following: hypertension, hypotension, heart rate, oxygen saturation, sleep, fatigue medication changes, seizure, headache/neck pain, fever, fainting, scalp/skin breakdown, tinnitus, dizziness, nausea, vomiting, confusion, and contraindicated substance use.
  Adverse event reporting logs were completed and reported to the IRB.
Arm/Group | Open Label iTBS+Yoga
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 3/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label iTBS+Yoga (N=19)
headache (Nervous system disorders) | 3 (3) — 3 individuals had headaches, resulting in 1 participant self-withdrawing. For this person, the headaches started ~3 days after the first session. This participant had a history of occasional unlocalized headaches.

LIMITATIONS AND CAVEATS:
The main limitations were the small sample size, open-label design, and lack of a control group. As this was a pilot we did not assess for multiple comparisons. Our satisfaction ratings and qualitative interviews assessing acceptability may be biased as they were only done for those completing all 6 intervention sessions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/04/NCT04517604/Prot_SAP_002.pdf
  • Informed Consent Form (2022-02-23): https://cdn.clinicaltrials.gov/large-docs/04/NCT04517604/ICF_003.pdf